CLINICAL TRIAL: NCT04438941
Title: Contribution of a Prone Team in Intensive Care During the Covid-19 Epidemic
Acronym: COVID-PRONE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7911
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Sars-CoV2
Keywords: Mechanical ventilation; ICU; Covid-19; SARS-CoV-2; ARDS
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-CoV-2 induced by COVID 19, involved the hospitalization of 101,932 patients in France, including 4,007 in intensive care (source: Santé Publique France). Alsace was one of the most affected regions on the metropolitan territory with a large number of patients hospitalized at the University Hospital of Strasbourg.

In view of the seriousness of the epidemic and the rapid arrival of new patients requiring mechanical ventilation, 3 new intensive care units have been created on the NHC site alone, making it possible to accommodate a maximum of 111 patients (compared to 52 during normal periods).

ELIGIBILITY:
Criteria for inclusion :

* Major patient (≥18 years old)
* Patient hospitalized in intensive care at the NHC, diagnosed COVID + and requiring a VD session of which at least one is performed by the dedicated team.
* patient who has not expressed, after information, his or her opposition to the re-use of his or her data for the purposes of this research

Exclusion criteria :

* Subject who expressed opposition to participating in the study
* Subject under guardianship, curatorship or safeguarding of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in intensive care at the NHC, diagnosed COVID + and requiring a VD session
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Analysis of the effect of prone position in patients with covid-19 in intensive care | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie-Réanimation - Nouvel Hôpital Civil, Strasbourg, France